CLINICAL TRIAL: NCT03945357
Title: Reducing INfection at the Surgical SitE With Antibiotic Irrigation During Ventral Hernia Repair (RINSE Trial)
Acronym: RINSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: The Cleveland Clinic (Other); Penn State University (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00087360
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Ventral Hernia Repair
Keywords: Infection; hernia repair
MeSH Terms: conditions — Infections | interventions — Gemcitabine; Clindamycin; Saline Solution

STUDY DESIGN:
Intervention Model Description: The study design would be a registry-based RCT through the AHSQC to evaluate the effect of dual antibiotic irrigation at the time of mesh placement during open RM +/-TAR OVHR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Saline Irrigation (Active Comparator): Normal saline is to be placed into the dissected retromuscular space AFTER placement and fixation of mesh. This should fill the cavity completely to the level of the skin. Irrigant is to be left to stand for a total of three minutes and then evacuated. Additional irrigation with saline PRIOR to the randomization is permitted at the surgeons' discretion for hemostasis with no requirement for duration. Additional saline irrigation of the subcutaneous space after fascia closure should be performed prior to skin closure.
  Interventions: Drug: Normal saline
- Antibiotic Irrigation (Active Comparator): Antibiotic solution is prepared consisting of 240 mg gentamicin and 600 mg clindamycin in 500 ml saline to ensure proper concentration. This solution should be placed into the dissected retromuscular space AFTER placement and fixation of mesh. This should fill the cavity completely to the level of the skin. Irrigant is to be left to stand for a total of three minutes and then evacuated. Additional irrigation with saline PRIOR to the randomization is permitted at the surgeons' discretion for hemostasis with no requirement for duration. Additional antibiotic irrigation of the subcutaneous space after fascia closure should be performed prior to skin closure. This second irrigation is not timed.
  Interventions: Drug: Gemcitabine/ clindamycin

INTERVENTIONS:
Drug: Gemcitabine/ clindamycin — Comparison of saline solution rinse vs antibiotic rinse
  Arms: Antibiotic Irrigation
Drug: Normal saline — Comparison of saline solution rinse vs antibiotic rinse
  Arms: Saline Irrigation

SUMMARY:
This is a study to determine if the incidence of infection at the Surgical SitE is impacted if with Antibiotic Irrigation is used during Ventral Hernia Repair (RINSE Trial)

DETAILED DESCRIPTION:
Surgical site infection (SSI) is common after open ventral hernia repair. Numerous factors contribute, including patient comorbidities, operative technique, and degree of contamination of the case. SSI often requires prolonged hospital length of stay (LOS), readmission, or other procedural intervention. One potential intervention to reduce SSI is the use of antibiotic irrigation, which has been shown to reduce SSI in colorectal surgery in a recent randomized control trial. We retrospectively evaluated our use of dual antibiotic irrigation at the time of mesh placement during open ventral hernia repair (OVHR), demonstrating a significant reduction in SSI (16.5 vs 5.4%) using a combination of gentamicin and clindamycin irrigation when compared to saline alone.

We plan to complete a registry-based, randomized clinical trial (RCT) through the Americas Hernia Society Quality Collaborative (AHSQC) to further assess the impact of dual antibiotic irrigation on SSI after OVHR with mesh. This will include patients undergoing open retromuscular (RM) repair with or without transversus abdominis myofascial advancement flap (TAR) with placement of permanent synthetic mesh (mid-weight, large-pore polypropylene). Power analysis based on only this subset of patients from our initial study indicates a total of 210 patients are needed to demonstrate a significant reduction in SSI using antibiotic irrigation vs saline irrigation alone.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 y/o.
* Elective, open ventral hernia repair in a retromuscular fashion, with or without TAR.
* Clean, clean-contaminated, or contaminated wounds.

Exclusion Criteria:

* Age <18 y/o.
* Pregnancy.
* Emergency hernia repair.
* Laparoscopic, robotic, or hybrid approach.
* Dirty wounds.
* Use of biologic or absorbable synthetic mesh.
* Onlay, intraperitoneal or preperitoneal mesh placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Warren, MD, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Prisma Health Upstate, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There will be no patient information shared

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saline Irrigation | Antibiotic Irrigation
Started | 124 | 126
Completed | 121 | 120
Not Completed | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline Irrigation | Antibiotic Irrigation | Total
Number analyzed (Participants) | 124 | 126 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 69 | 127
  >=65 years | 66 | 57 | 123
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 61 | 135
  Male | 50 | 65 | 115
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Surgical Site Infection
Description: Number of participants with Surgical Site Infections
Time Frame: 30 days
Population: 111 subjects in the saline group reached the 30 day visit. 110 subjects in the antibiotic group reached the 30 day visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Saline Irrigation | Antibiotic Irrigation
Number analyzed (Participants) | 111 | 110
Participants | 11 | 10

2. Secondary Outcome: Incidence of SSI Requiring Intervention
Description: Number of participants with SSI requiring reoperation or other procedural intervention at 30 days.
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Saline Irrigation | Antibiotic Irrigation
Number analyzed (Participants) | 111 | 110
Participants | 8 | 8

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Saline Irrigation | Antibiotic Irrigation
All-Cause Mortality (participants affected / at risk) | 1/124 | 3/126
Serious Adverse Events (participants affected / at risk) | 9/124 | 5/126
Other Adverse Events (participants affected / at risk) | 13/124 | 7/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saline Irrigation (N=124) | Antibiotic Irrigation (N=126)
bowel obstruction (Gastrointestinal disorders) | 1 | 1
hematoma (Blood and lymphatic system disorders) | 2 | 0
respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 | 3
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
alcohol withdrawal (Injury, poisoning and procedural complications) | 1 | 0
ascites (Gastrointestinal disorders) | 1 | 0
wound infection (Infections and infestations) | 1 | 0
lethargy (General disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saline Irrigation (N=124) | Antibiotic Irrigation (N=126)
ileus (Gastrointestinal disorders) | 13 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT03945357/Prot_SAP_001.pdf